CLINICAL TRIAL: NCT05820971
Title: Impact of a Short Form of the CONSORT Checklist for Peer Reviewers to Improve the Reporting of Randomised Controlled Trials Published in Biomedical Journals: a Randomised Controlled Trial
Brief Title: A Short CONSORT Checklist for Peer Reviewers to Improve the Reporting of Randomised Controlled Trials Published
Acronym: CONSORT-PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CONSORT-PR 2019; R62779/RE001 (Other: MEDICAL SCIENCES INTERDIVISIONAL RESEARCH ETHICS COMMITTEE, University of Oxford); P300PB_177933 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2019-05-23; First posted 2023-04-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2019-05

CONDITIONS: Adequate Reporting in Randomized Controlled Trials

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-short plus usual practice (Experimental): After accepting to review an article, peer reviewers will receive the automated, journal specific standard email with general information as per each journal's usual practice (e.g. where to access the manuscript, date when the peer review report is due). In addition, peer-reviewers who received a manuscript which was randomised to C-short will receive an additional email including a short version of the CONSORT checklist together with a short explanation of those items.
  Interventions: Other: C-short plus usual practice
- Usual practice (No Intervention): After accepting to review an article, peer reviewers will receive the automated, journal specific standard email with general information as per each journal's usual practice.

INTERVENTIONS:
Other: C-short plus usual practice — Peer reviewer will be reminded of the following 10 CONSORT items (including a short description):
  * Outcomes (6a)
  * Sample size (7a)
  * Sequence generation (8a)
  * Allocation concealment (9)
  * Blinding (11a)
  * Outcomes and estimation (17a/b)
  * Harms (19)
  * Registration (23)
  * Protocol (24)
  * Funding (25)
  Arms: C-short plus usual practice

SUMMARY:
Transparent and accurate reporting is key, so that readers can adequately interpreting the results of a study. Despite improvement with implementation of the CONSORT Statement (CONsolidated Standards for Reporting Trials), there remain major reporting deficiencies in published randomized controlled trials (RCT). The aim of this project is to evaluate whether reminding peer reviewers of the most important CONSORT items (including a short explanation of those items) will result in higher adherence to CONSORT guidelines in published RCTs. During the standard peer-review process, peer-reviewers will be randomly allocated to use either (i) a short version of the CONSORT checklist including the ten most important and poorly reported CONSORT items as defined by a group of experts of the CONSORT Statement (C-short); or (ii) no checklist. The aim is to find an intervention which improves the reporting, making it easier for readers to adequately interpret the presented results.

DETAILED DESCRIPTION:
The CONSORT Statement (CONsolidated Standards for Reporting Trials), is perhaps the most important reporting guideline designed to help improve the transparency and quality of reporting of randomized controlled trials. Despite some improvement in reporting following the implementation of the CONSORT Statement, there still remain major reporting deficiencies in published RCTs. The investigators are conducting a multicentre randomized controlled trial to evaluate whether reminding peer reviewers of the most important CONSORT items (including a short explanation of those items) will result in higher adherence to CONSORT guidelines in published RCTs. During the standard peer-review process, peer-reviewers will be randomly allocated to use either (i) a short version of the CONSORT checklist including the ten most important and poorly reported CONSORT items as defined by a group of experts of the CONSORT Statement (C-short plus usual practice); or (ii) no checklist (usual practice). The primary outcome of this study will be the difference of the mean proportion of adequately reported items of the 10 most important and poorly reported CONSORT items between the two intervention arms.

The Full protocol is available on Open Science Framework where the study was prospectively registered (https://osf.io/c4hn8)

ELIGIBILITY:
Inclusion Criteria:

* Included journals must:
* Endorse the CONSORT Statement (e.g. assessed via journals Instruction to Authors);
* Publish primary results of at least five RCTs in 2017 (identified in a brief PubMed search as publishing RCTs in 2017)

Included Manuscript must:

-Report primary results of an RCTs for which the journal decides to send out for external peer review (since the 10 chosen CONSORT checklist items are applicable to different study designs, the investigators will include all RCTs regardless of study design [e.g. parallel group trial, cluster trial, superiority trial, non-inferiority trial]).

Exclusion Criteria:

* Articles presenting clearly secondary trial results.
* Articles presenting clearly additional time points and not the time point where the primary result was measured.
* Economic analyses
* Any other analyses derived from an RCT dataset not including the study's main results -- -RCTs which are clearly labelled as a pilot or feasibility study
* RCTs randomising animals or cells instead of individuals

Included peer-reviewers:

-Peer reviewers that were invited following usual journal practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Completeness of reporting | Through study completion, an average of 1 year
  The primary outcome of this study will be the difference of the mean proportion of adequately reported items of the 10 most important and poorly reported CONSORT items between the two intervention arms.

SECONDARY OUTCOMES:
Completeness of reporting | Through study completion, an average of 1 year
  Mean proportion of adequate reporting of the 10 most important and poorly reported CONSORT items, considering each sub-item (see also "Assessment of outcomes") as a separate item.
Completeness of reporting | Through study completion, an average of 1 year
  Mean proportion for each of the 10 most important and poorly reported CONSORT items separately (including also separate analysis of sub-items).
Time from assigning an academic editor until the first decision (as communicated to the author after the first round of peer-review). | Through study completion, an average of 4 months; will be assessed from routinely collected data
Proportion of articles directly rejected after the first round of peer-review | Through study completion, an average of 4 months; will be assessed from routinely collected data
Proportion of articles published | Through study completion, an average of 9 months; will be assessed from routinely collected data

OTHER OUTCOMES:
Peer reviewer comments for any reference to CONSORT and trial reporting | Assessed from available peer-reviewer responses; on average 3 months after randomisation
  For journals where peer reviewer comments are subsequently published alongside the published article, the investigators will examine the peer reviewer comments for any reference to CONSORT and trial reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Hopewell, Ass. Prof, Study Chair — Centre for Statistics in Medicine, Oxford University
Locations (2):
- Public Library of Science (PLOS), San Francisco, California, United States
- The BMJ Publishing Group, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish the anonymised data set together with the main publication.
Supporting Information: Study Protocol
Time Frame: The investigators plan to submit the study protocol to a peer reviewed journal in 2019.
URL: https://bmjopen.bmj.com/content/10/3/e035114.long

REFERENCES:
- [Derived] Speich B, Mann E, Schonenberger CM, Mellor K, Griessbach AN, Dhiman P, Gandhi P, Lohner S, Agarwal A, Odutayo A, Puebla I, Clark A, Chan AW, Schlussel MM, Ravaud P, Moher D, Briel M, Boutron I, Schroter S, Hopewell S. Reminding Peer Reviewers of Reporting Guideline Items to Improve Completeness in Published Articles: Primary Results of 2 Randomized Trials. JAMA Netw Open. 2023 Jun 1;6(6):e2317651. doi: 10.1001/jamanetworkopen.2023.17651. PMID 37294569